CLINICAL TRIAL: NCT00261794
Title: Computer Assisted Cognitive Remediation for Schizophrenia
Brief Title: Cognitive Remediation for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bellack, Alan - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: D3153R
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Schizophrenia
Keywords: cognition; schizophrenia; treatment
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): computer-assisted cognitive remediation (CACR)
  Interventions: Behavioral: computer-assisted cognitive remediation (CACR)
- 2 (Active Comparator): computer-based cognitive activity
  Interventions: Behavioral: manualized computer control condition (RC).

INTERVENTIONS:
Behavioral: computer-assisted cognitive remediation (CACR) — 36 individual computer sessions with a staff clinician. computer activities consist of commercially available educational software designed for use in the classroom.
  Other Names: CACR
  Arms: 1
Behavioral: manualized computer control condition (RC). — 36 sessions of a manualized computer control condition.
  Other Names: RC
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of an innovative, computer driven cognitive rehabilitation program for unemployed veterans with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia leads to a striking array of negative outcomes, including profound deficits in the ability to fulfill desired and expected community roles. Chronic under employment and unemployment are among the most serious of these consequences. VA treats over 100,000 veterans with schizophrenia spectrum disorders, the majority of whom are unable to work competitively and do not participate in VA vocational rehabilitation programs despite the fact that VA is committed to enhancing the ability of these veterans to work. Within VA, a major vehicle for helping veterans to become employed is the Compensated Work Therapy (CWT) program, yet in FY2001 only 800 of the roughly 14000 veterans treated in CWT had SMI diagnoses, and only a subset of those 800 had schizophrenia. A number of factors contribute to low participation in vocational rehabilitation and poor work outcomes, but recent data suggest that one of the most important is cognitive impairment. People with schizophrenia have significant deficits in multiple areas of neurocognition, including secondary and working memory, attention, and executive functioning. These impairments have been shown to play a major role in functional outcome, including the ability to benefit from rehabilitation and to work. As a result, there has been increasing interest in the potential for improving neurocognitive functioning via cognitive rehabilitation. While several programs have yielded promising data, currently there is no empirically validated approach.The purpose of this project is to evaluate the efficacy of an innovative, computer driven cognitive rehabilitation program we have developed: Computer Assisted Cognitive Remediation (CACR). Veterans with schizophrenia who are unemployed and not participating in vocational rehabilitation will be recruited and randomly assigned to one of two conditions: a) 36 sessions of CACR; or b) 36 sessions of a manualized computer control condition (RC). The efficacy of CACR will be assessed on a range of outcome domains, including neuropsychological test, measures of every day and social problem solving, self-reported cognitive functioning and self-efficacy, and work readiness. All subjects will be referred to CWT at the conclusion of treatment and we will assess how many receive work assignments, and work performance (over 3-months) of those who begin work. We hypothesize that CACR will be more effective than the control treatment in each domain.The results of this project could have important implications for treatment of veterans with schizophrenia. CACR is a manualized program that can be administered by BA level staff. If demonstrated to be efficacious, it could be disseminated throughout VA and have a beneficial impact on vocational outcomes and the quality of life of veterans with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Current DSM-IV diagnoses of schizophrenia or schizoaffective disorder
2. Stable clinical course and antipsychotic treatment on a new generation antipsychotic other than clozapine and/or a dose of first generation antipsychotic equivalent to 10 mg. or less of haloperidol for one month prior to enrollment
3. Age between 18 and 64 years
4. Voluntary consent after receiving full information about the study

Exclusion Criteria:

1. Documented history of neurological disorder or significant head trauma with extended loss of consciousness
2. Physical limitations (e.g., with hearing or vision) that would interfere substantially with the use of computer-based exercises
3. Current treatment with a first generation antipsychotic medication at a dose equivalent to more than 10 mg. of haloperidol
4. Current treatment with benztropine mesylate at a daily does greater than 4 mg
5. Current treatment with trihexyphenidyl at a daily dose greater than 15 mg
6. Current treatment that combines benztropine mesylate with trihexyphenidyl
7. Current treatment with diphenhydramine
8. Current competitive employment or participation (current or within past 3 months) in a program designed to secure competitive employment (e.g., CWT)
9. Mini Mental Status Examination (MMSE) score of less than 23
10. Diagnosis of current Substance Dependence according to DSM-IV criteria

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
cognitive performance and every day problem solving | post-treatment and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Bellack, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Bellack AS, Gold JM, Buchanan RW. Cognitive rehabilitation for schizophrenia: problems, prospects, and strategies. Schizophr Bull. 1999;25(2):257-74. doi: 10.1093/oxfordjournals.schbul.a033377. PMID 10416730
- [Result] Bellack AS. Skills training for people with severe mental illness. Psychiatr Rehabil J. 2004 Spring;27(4):375-91. doi: 10.2975/27.2004.375.391. PMID 15222149
- [Result] Dickinson D, Tenhula W, Morris S, Brown C, Peer J, Spencer K, Li L, Gold JM, Bellack AS. A randomized, controlled trial of computer-assisted cognitive remediation for schizophrenia. Am J Psychiatry. 2010 Feb;167(2):170-80. doi: 10.1176/appi.ajp.2009.09020264. Epub 2009 Dec 15. PMID 20008941